CLINICAL TRIAL: NCT04380727
Title: Almitrine and Severe COVID-19 Patients in ICU [Almitrine et Patients COVID-19 en Reanimation (French)]
Brief Title: Almitrine and COVID-19 Related Hypoxemia
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI080_2
Record Dates: First submitted 2020-04-28; First posted 2020-05-08 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Hypoxic Respiratory Failure
Keywords: Hypoxic pulmonary vasoconstriction; Prone position; intra-pulmonary shunt; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Almitrine: Administration of 4 mcg/kg/min iv almitrine bismesylate (Vectarion®, Servier Laboratory, France), over 30-45 min followed by 12 mcg/kg/min infusion rate. Because of a shortage of drug store at national level, a protocol using continuous infusion was not considered. Some patients may receive the drug for 36 hours depending on availability..
- Control: To eliminate the eventuality of a spontaneous evolution of hypoxia, these patients were matched to control COVID-19 patients treated without almitrine (time control).

SUMMARY:
In severe COVID-19 pulmonary failure, the profound hypoxemia is mainly related to pulmonary vasodilation with altered hypoxic pulmonary vasoconstriction (HPV). Besides prone positioning, other non-ventilatory strategies may reduce the intrapulmonary shunt. This study has investigated almitrine, a pharmacological option used in standard care to improve oxygenation.

A case control series of mechanically ventilated confirmed COVID-19 patients was recorded.

At stable ventilatory settings, consecutive patients received two doses of almitrine (4 and 12 mcg/kg/min) at 30-45 min interval each, and were compared to 7 "control" COVID-matched patients conventionally treated.

The end-point was the reduction of intra-pulmonary shunt, with an increase in partial pressure of arterial oxygen (PaO2) and central venous oxygen saturation (ScvO2).

DETAILED DESCRIPTION:
The clinical presentation of COVID-19 disease is heterogenous, ranging from no symptoms to severe acute respiratory failure (ARF), which may have a poor prognosis. A severe hypoxemia is associated with preserved respiratory mechanical properties, in particular the pulmonary system compliance.

The hypoxia during the early phase seems to mainly result from an important ventilation/perfusion (VA/Q) mismatch associated with an altered pulmonary vasoconstriction. The "protective" mechanism called hypoxic pulmonary vasoconstriction (HPV) normally reduces the blood flow in poorly or non-ventilated areas towards aerated zones leading to reduce the (VA/Q) mismatch. HPV seems poorly functional in COVID-19 severe patients in absence of "cor pulmonale".

According to the French National agency for Drug Security (ANSM, Paris, France), only iv almitrine is indicated for hypoxic acute respiratory failure as Drug of Major Therapeutic Interest. This molecule is a routine option in the treatment strategy of severe hypoxemia.

The investigators studied COVID-19 patients mechanically ventilated at FiO2 1 with a severe intrapulmonary shunt during their early phase. The emergency conditions and the acute high inflow of patients to ICU impeded the design of a randomized control trial. To eliminate the eventuality of a spontaneous evolution of hypoxia, these patients will be compared with control-matched COVID patients treated conventionally.

ELIGIBILITY:
Inclusion Criteria :

* a positive RT- PCR,
* a highly suggestive thoracic CTScan, and
* a severe hypoxemia leading to intubation for less than 3 days
* mechanically ventilated at FiO2 1 with a severe intrapulmonary shunt during their early phase

Group : patient who has been treated with almitrine (4 mcg/kg/min iv almitrine bismesylate (Vectarion®, Servier Laboratory, France) then 12 mcg/kg/min infusion rate) during their hospital treatment.

Control group : Matched COVID-19 patients, on gender, age, BMI and duration of mechanical ventilation, with serial measurements corresponding to the duration of almitrine testing (8 hours), with same inclusion and exclusion criteria.

Exclusion Criteria:

* the presence of an acute cor-pulmonale on the trans-thoracic 2D Echo-Doppler
* abnormal liver function tests
* hyperlactatemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between March16 and April 20, 2020, COVID-19 patients referred to ICU age, gender, BMI, Hb The recorded parameters were: the ventilatory settings unchanged along the protocol, including FiO2, PEEP level, tidal volume (VT), peak inspiratory pressure, plateau pressure; haemoglobin concentration, blood gases simultaneously sampled on the arterial catheter and on the central catheter to assess central venous oxygen saturation SvcO2, and arterial lactate, right atrial pressure; cardiac output when possible (Mostcare®, Vygon, Ecouen, France).
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Changes from baseline PaO2 (mmHg) | 45 minutes after almitrine infusion
  Partial pressure of oxygen in arterial blood
Changes from baseline ScvO2 (%) | baseline and 45 minutes after almitrine infusion
  central venous oxygen saturation

SECONDARY OUTCOMES:
Changes from baseline PaO2 (mmHg) | 8 hours
  partial pressure of oxygen in arterial blood
Changes from baseline ScvO2 (%) | 8 hours
  central venous oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Marie Reine LOSSER, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Universitaire NANCY, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided
Collaborative register on COVID-19 having benn treated with almitrine

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Gattinoni L, Coppola S, Cressoni M, Busana M, Rossi S, Chiumello D. COVID-19 Does Not Lead to a "Typical" Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2020 May 15;201(10):1299-1300. doi: 10.1164/rccm.202003-0817LE. No abstract available. PMID 32228035
- [Background] Payen DM, Gatecel C, Plaisance P. Almitrine effect on nitric oxide inhalation in adult respiratory distress syndrome. Lancet. 1993 Jun 26;341(8861):1664. doi: 10.1016/0140-6736(93)90801-m. No abstract available. PMID 8100027
- [Background] B'chir A, Mebazaa A, Losser MR, Romieu M, Payen D. Intravenous almitrine bismesylate reversibly induces lactic acidosis and hepatic dysfunction in patients with acute lung injury. Anesthesiology. 1998 Oct;89(4):823-30. doi: 10.1097/00000542-199810000-00005. PMID 9777998